CLINICAL TRIAL: NCT07129499
Title: A Multicenter, Randomized, Double-blind, Placebo-Controlled Clinical Trial of Shenbai Granules for Preventing Malignant Transformation of High-Risk Colorectal Adenomas
Brief Title: Shenbai Granules for Preventing Malignant Transformation of High-risk Colorectal Adenomas
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangsu Famous Medical Technology Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); First Affiliated Hospital of Harbin Medical University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The Second Affiliated Hospital of Chongqing Medical University (Other); Chongqing Traditional Chinese Medicine Hospital (Other); The Second Hospital of Shandong University (Other); Shengjing Hospital (Other); Shenzhen Hospital of Southern Medical University (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Sichuan Provincial People's Hospital (Other); Shanxi Provincial People's Hospital (Other Government); Affiliated Hospital of Nanjing University of Chinese Medicine (Other); RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024ZD0520804
Record Dates: First submitted 2025-08-07; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Adenoma; High Risk; TCM
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shenbai Granules (Experimental): Shenbai Granules is a traditional Chinese medicine preparation formulated from eight herbal ingredients, including Sophorae Flavescentis Radix (Kushen), Coptidis Rhizoma (Huanglian), and other herbs. It exerts therapeutic effects by clearing heat and drying dampness, while simultaneously invigorating the spleen and replenishing qi.
  Interventions: Drug: Shenbai Granules
- Placebo (Placebo Comparator): The placebo was formulated using Shenbai Granules dry extract powder at 2% (w/w) of the equivalent dose found in the compound herbal granules, supplemented with colorants and flavoring agents to ensure visual and gustatory consistency with the Shenbai Granules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Shenbai Granules — 10 g/bag, two bags each time, twice a day, monthly for 30 days for 6 months.
  Other Names: Treatment group
  Arms: Shenbai Granules
Drug: Placebo — 10 g/bag, two bags each time, twice a day, monthly for 30 days for 6 months.
  Other Names: Control group
  Arms: Placebo

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled trial will enroll 450 patients with completely resected high-risk colorectal adenoma (HR-CRA), randomly assigned (1:1) to 6 months of Shenbai Granules (SBG) or placebo, followed for 3 years post-polypectomy. Primary endpoint: 3-year cumulative incidence of metachronous HR-CRA. Secondary endpoints: incidence, number, size, distribution, histology of low-risk adenomas and serrated lesions, and colorectal cancer occurrence.

DETAILED DESCRIPTION:
High-risk colorectal adenomas (HR-CRAs) are a recognized precursor lesion for colorectal cancer, with 25-40% of patients developing metachronous adenomas within 3 years after endoscopic resection. Low-dose aspirin is the only agent supported by high-level evidence for reducing the incidence of metachronous HR-CRAs, but its use is limited by bleeding risks. Although previous studies on the traditional Chinese medicine compound Shenbai Granules (SBG) have suggested its potential in preventing metachronous HR-CRAs, sufficient evidence from randomised controlled trials (RCTs) is still lacking. This trial aims to confirm the efficacy and safety of SBG in preventing the development of metachronous adenomas and subsequent carcinogenesis, and to identify clinical predictors of treatment response to define the optimal target population. This multicentre, randomised, double-blind, placebo-controlled trial will enroll 450 patients with endoscopically resected HR-CRAs. Participants will be randomly allocated 1:1 to receive either SBG (n=225) or a matching placebo (n=225). The trial comprises a 14-day screening period, a 6-month treatment phase, and a 30-month surveillance phase, including four on-site visits and one telephone follow-up. The primary endpoint is the three-year cumulative incidence of metachronous HR-CRA. Secondary endpoints include the incidence of metachronous low-risk adenomas and serrated lesions within the same 3-year window, cumulative number and size of lesions, anatomic distribution, histopathology, and the incidence of colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

All of the following criteria must be met for enrolment:

1. Aged 40-75 years, regardless of gender;
2. High-quality colonoscopy performed within 14 days before randomisation, with initial endoscopic resection of all polyps and histological confirmation of at least one HR-CRA criteria;
3. Complete endoscopic resection of every detected lesion;
4. TCM syndrome differentiation of "spleen deficiency with dampness-heat";
5. Signed informed consent and willingness to comply with long-term follow-up. a: High-quality colonoscopy criteria: Boston Bowel Preparation Scale score ≥ 6, cecal intubation confirmed by visualization of the ileocecal valve, and withdrawal time (excluding biopsy and polypectomy) ≥ 6 minutes.

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from the trial:

1. Concomitant malignancy or history of malignancy in the digestive system;
2. Personal or family history of familial adenomatous polyposis or hereditary non-polyposis colorectal cancer (Lynch syndrome);
3. History of inflammatory bowel disease;
4. Malignancy in any other organ system within 5 years before screening, except for adequately treated thyroid carcinoma, cervical carcinoma in situ, basal or squamous cell skin carcinoma, or ductal carcinoma in situ of the breast cured by radical surgery;
5. Clinically significant organic disorders or neuro-psychiatric conditions that may affect treatment or prognosis, including but not limited to severe cardiovascular or cerebrovascular disease, autoimmune disease, motor, haematological, gastrointestinal, respiratory, immune, circulatory, reproductive, genitourinary, or endocrine disorders; coagulation abnormalities; or serious post-procedural complications (e.g., gastrointestinal bleeding, perforation, cholangitis, intra-abdominal infection, cardiorespiratory depression, mesenteric tear, or pneumoperitoneum), serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.5 × the upper limit of normal (ULN), or alkaline phosphatase (ALP) >2 × ULN;
6. Active gastrointestinal disease, conditions predisposing to perforation, or disorders that could substantially interfere with the absorption, distribution, metabolism, or excretion of the investigational drug, such as inability to take oral medication, uncontrolled nausea or vomiting, intestinal obstruction, or chronic diarrhoea;
7. Within 3 months before screening, continuous use for ≥3 months of ≥2 doses per week (with <2-week interruption) of agents potentially protective against colorectal adenoma: NSAIDs (e.g., aspirin, ibuprofen, celecoxib), metformin, berberine hydrochloride, folic acid, vitamin D, selenium, calcium, systemic immunotherapy, or Chinese patent medicines or decoctions labelled for "tonifying spleen and augmenting qi, clearing heat and eliminating dampness". Subjects may be enrolled after a washout of 1 month or ≥5 drug half-lives, whichever is longer;
8. Cold-pattern manifestations such as aversion to cold, cold pain in the waist/abdomen, cold extremities, or preference for hot drinks;
9. Pregnant or lactating women, or men and women of child-bearing potential with plans to conceive during the trial or within 7 months after trial completion;
10. Participation in another drug or device trial within 1 month or < 5 half-lives of the investigational agent (whichever is longer) before screening, concurrent participation in another trial, or intention to participate in any other clinical trial during this trial;
11. Known allergy or hypersensitivity to ≥ 2 drugs or foods, or hypersensitivity to any component of the trial medication;
12. Any other condition that, in the opinion of the investigator, makes the subject unsuitable for enrolment (e.g., poor expected compliance, cognitive impairment).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative detection rate of metachronous high-risk colorectal adenomas within 3 years after the first dose. | 1, 3 years
  The proportion of patients found to have metachronous high-risk colorectal adenomas during surveillance colonoscopy within 3 years after baseline adenoma resection. Colonoscopy will be performed in the first and third years.

SECONDARY OUTCOMES:
Cumulative detection rate of metachronous low-risk colorectal adenomas within 3 years after the first dose. | 1, 3 years
  The proportion of patients found to have metachronous low-risk colorectal adenomas during surveillance colonoscopy within 3 years after baseline adenoma resection. Colonoscopy will be performed in the first and third years.
Cumulative counts of metachronous colorectal adenomas detected within 3 years after the first dose. | 1, 3 years
  The cumulative counts of metachronous colorectal adenomas detected during colonoscopic surveillance within 3 years after baseline adenoma resection. Colonoscopy will be performed in the first and third years.
The average number of metachronous colorectal adenomas detected within 3 years after the first dose. | 1, 3 years
  The average number of metachronous colorectal adenomas detected during colonoscopic surveillance within 3 years after baseline adenoma resection. Colonoscopy will be performed in the first and third years.
Size of metachronous colorectal adenomas detected within 3 years after the first dose. | 1, 3 years
  The average size of metachronous colorectal adenomas detected during colonoscopic surveillance within 3 years after baseline adenoma resection. Colonoscopy will be performed in the first and third years.
Location of metachronous colorectal adenomas detected within 3 years after the first dose. | 1, 3 years
  The location (left colon, right colon, rectum) of metachronous colorectal adenomas detected during colonoscopic surveillance within 3 years after baseline adenoma resection. Colonoscopy will be performed in the first and third years.
Pathology of metachronous colorectal adenomas detected within 3 years after the first dose. | 1, 3 years
  The pathological types (histological architecture: tubular adenoma, villous adenoma, tubulovillous adenoma; and degree of dysplasia: high-grade intraepithelial neoplasia, low-grade intraepithelial neoplasia) of metachronous colorectal adenomas detected during colonoscopic surveillance within 3 years after baseline adenoma resection. Colonoscopy will be performed in the first and third years.
Cumulative detection rate of serrated lesions within 3 years after the first dose. | 1, 3 years
  The proportion of cases with serrated lesions identified during colonoscopy surveillance within 3 years after baseline adenoma resection, relative to the total number of cases in the cohort. Colonoscopy will be performed in the first and third years.
Cumulative incidence of serrated lesions detected within 3 years after the first dose. | 1, 3 years
  The cumulative incidence of serrated lesions detected during colonoscopic surveillance within 3 years after baseline adenoma resection. Colonoscopy will be performed in the first and third years.
The average number of serrated lesions detected within 3 years after the first dose. | 1, 3 years
  The average number of serrated lesions detected during colonoscopic surveillance within 3 years after baseline adenoma resection. Colonoscopy will be performed in the first and third years.
Size of serrated lesions detected within 3 years after the first dose. | 1, 3 years
  The average size of serrated lesions detected during colonoscopic surveillance within 3 years after baseline adenoma resection. Colonoscopy will be performed in the first and third years.
Location of serrated lesions detected within 3 years after the first dose. | 1, 3 years
  The location distribution (left colon, right colon, rectum) of serrated lesions detected during colonoscopic surveillance within 3 years after baseline adenoma resection. Colonoscopy will be performed in the first and third years.
Pathological types of all serrated lesions detected within 3 years after the first dose. | 1, 3 years
  The pathological types (colorectal serrated lesion, sessile serrated lesion, hyperplastic polyp) of serrated lesions will be detected during colonoscopic surveillance within 3 years after baseline adenoma resection. Colonoscopy will be performed in the first and third years.
Incidence of colorectal cancer within 3 years after the first dose. | 1, 3 years
  The proportion of cases with interval colorectal cancer detected during surveillance colonoscopy within 3 years after baseline adenoma resection, relative to the total number of cases in the cohort. Colonoscopy will be performed in the first and third years.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Nanjing University of Chinese Medicine, Nanjing, Jiangsu, China